CLINICAL TRIAL: NCT00112983
Title: TRIUMPH: A Hemoglobin Stabilization and Transfusion Reduction Efficacy and Safety Clinical Investigation, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Using Eculizumab in Paroxysmal Nocturnal Hemoglobinuria Patients
Brief Title: Eculizumab in Treating Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: ALEXION-C04-001; UCLA-0406101-01; CDR0000409569 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2005-06

CONDITIONS: Leukemia
Keywords: adult acute lymphoblastic leukemia; adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — eculizumab

INTERVENTIONS:
Biological: eculizumab

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of eculizumab may prevent leukemia and stop the destruction of red blood cells in patients with paroxysmal nocturnal hemoglobinuria.

PURPOSE: This randomized phase III trial is studying how well eculizumab works in treating patients with paroxysmal nocturnal hemoglobinuria.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of eculizumab in patients with transfusion-dependent hemolytic paroxysmal nocturnal hemoglobinuria.
* Determine the efficacy of this drug, in terms of hemoglobin stabilization and the number of packed red blood cell units transfused during the 26-week treatment period, in these patients.

Secondary

* Compare the occurrence of transfusion avoidance, hemolysis (measured by lactate dehydrogenase [LDH] area under the curve), and the changes in fatigue during the 26-week treatment period in patients treated with this drug vs placebo.
* Compare LDH changes, quality of life changes, thrombosis, platelet activity, nitric oxide, and free hemoglobin measures during the 26-week treatment period in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to the number of packed red blood cell (PRBC) units transfused 1 year prior to screening (< 15 units vs 15-25 units vs > 25 units). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Within 10 days after PRBC transfusion (administered during the study observation period), patients receive placebo IV over 30 minutes once a week for 5 weeks and then once every 2 weeks for 21 weeks.
* Arm II: Within 10 days after PRBC transfusion (administered during the study observation period), patients receive eculizumab IV over 30 minutes once a week for 5 weeks and then once every 2 weeks for 21 weeks.

Quality of life is assessed at baseline; at weeks 0-4, 12, 20, and 26 during study treatment; then at weeks 1, 2, 4, and 8 after completion of study treatment.

After completion of study treatment, patients are followed at weeks 1, 2, 4, and 8.

PROJECTED ACCRUAL: Approximately 75 patients (37 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of paroxysmal nocturnal hemoglobinuria
* Must have required ≥ 4 episodes of transfusions for anemia or anemia-related symptoms within the past year

  * Mean pre-transfusion hemoglobin ≤ 10. 5 g/dL over the past year
* Glycosylphosphatidylinositol (GPI)-deficient red blood cell clone (type III cells) of ≥ 10% by flow cytometry
* Must have received 1 packed red blood cell transfusion during the study observation period (within 48 hours of the hemoglobin level that precipitated the transfusion) and within 1.5 g/dL of the mean pre-transfusion hemoglobin level over the past year

  * Pre-transfusion hemoglobin ≤ 9 g/dL with symptoms
  * Pre-transfusion hemoglobin ≤ 7 g/dL without symptoms
* Received Neisseria meningitidis vaccination at least 2 weeks before initiation of study therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count > 500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Lactate dehydrogenase ≥ 1.5 times upper limit of normal

Renal

* Not specified

Immunologic

* No known or suspected active bacterial infection
* No recurrent bacterial infections
* No history of meningococcal disease

Other

* No known or suspected hereditary complement deficiency
* No other condition that would increase the patient's risk or confound the outcome of the study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior bone marrow transplantation
* Concurrent epoetin alfa allowed*

Chemotherapy

* Not specified

Endocrine therapy

* Concurrent corticosteroids allowed**

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 30 days since prior participation in another investigational drug trial
* More than 30 days since prior investigational agents, devices, or procedures
* Concurrent immunosuppressants allowed*
* Concurrent warfarin allowed provided INR level is stable for the past 4 weeks and expected to remain stable during observation and study treatment
* Concurrent iron supplements or folic acid allowed**
* Concurrent low-molecular weight heparin allowed** NOTE: *Provided dose is stable for the past 26 weeks and during study observation and treatment

NOTE: **Provided dose is stable for the past 4 weeks and expected to remain stable (or decrease for corticosteroids) during study observation and treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Paquette, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States